CLINICAL TRIAL: NCT03400514
Title: A Retrospective, Self - Controlled, Single - Center Clinical Concordance Study Between Watson for Oncology and Clinician Practice
Brief Title: Clinical Concordance Study Between Watson for Oncology and Clinician Practice
Acronym: W001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Xiaochun Zhang, Professor, Qingdao University
Other Study IDs: XCZhang001
Record Dates: First submitted 2017-12-21; First posted 2018-01-17 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Artificial Intelligence
Keywords: Artificial intelligence; concordance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present, Watson for Oncology has been applied in 14 countries worldwide, including China, the United States, Holland, Thailand, India, Korea, Poland, Slovakia and Bangladesh. In a double-blind study involving 362 patients in India, treatment recommendations from Watson for Oncology (WFO) performed a high degree of consistency with their multidisciplinary tumor board. The investigators would recruit cancer patients diagnosed as lung cancer, breast cancer, gastric cancer, colon cancer， rectal cancer，cervical cancer or ovarian cancer according to the criteria of Watson for Oncology ，using the updated version of Watson for Oncology to explore the concordance of therapeutic regimen between WFO and physicians in the Affiliated Hospital of Qingdao University.

DETAILED DESCRIPTION:
This study was approved by the Affiliated Hospital of Qingdao University ethics committee.The investigators would randomly selected cancer patients, including lung cancer, breast cancer, gastric cancer, colon cancer，rectal cancer，cervical cancer and ovarian cancer patients, from the Affiliated Hospital of Qingdao University database according to the criteria of Watson for Oncology(supplementary materials). Case data would be extracted and input into the Watson system. WFO provided therapeutic recommendations in three categories: recommended, for consideration, and not recommended. Data would be analyzed retrospectively to compare the WFO's recommendations and actual therapeutic regimen in the hospital. Some actual regimen applications that were not available in WFO will be defined as "physician's choice". Overall, physician's recommendations would be defined as concordant with WFO if they corresponded to the recommended or consideration categories and as non-concordant if they corresponded to the not recommended or not available categories.

ELIGIBILITY:
Inclusion Criteria:

* a histology of lung cancer,breast cancer,gastric cancer, colon cancer， rectal cancer，cervical cancer and ovarian cancer
* had no prior systemic therapy and need neoadjuvant/adjuvant or metastatic therapy
* had prior neoadjuvant therapy, adjuvant therapy and/or surgery and are now metastatic
* have had prior surgery and now need adjuvant therapy
* seeking an additional therapy whose cancer has progressed beyond its initial metastatic therapy (second line)

Exclusion Criteria:

* not have confirmed diagnoses of invasive cancer
* under 18 years of age
* pregnant
* with multiple concurrent primary cancers or a local recurrence or a new primary at the same site of a previously treated cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients from outpatient and inpatient in our hospital
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
concordance | Day 0
  the concordance of therapeutic regimen between WFO and physicians in the Affiliated Hospital of Qingdao University

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zhang, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

REFERENCES:
- [Derived] Zhou N, Zhang CT, Lv HY, Hao CX, Li TJ, Zhu JJ, Zhu H, Jiang M, Liu KW, Hou HL, Liu D, Li AQ, Zhang GQ, Tian ZB, Zhang XC. Concordance Study Between IBM Watson for Oncology and Clinical Practice for Patients with Cancer in China. Oncologist. 2019 Jun;24(6):812-819. doi: 10.1634/theoncologist.2018-0255. Epub 2018 Sep 4. PMID 30181315